CLINICAL TRIAL: NCT05431426
Title: Open-label, Non-randomised, Parallel-group Study to Investigate the Pharmacokinetics, Safety and Tolerability Following Single Administration of CHF6001 in Subjects With Mild, Moderate and Severe Renal Impairment in Comparison With Matched Healthy Control Subjects
Brief Title: PK of CHF6001 in Subjects With Mild, Moderate and Severe Renal Impairment vs. Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLI-06001AA1-07; 2021-005567-43 (EudraCT Number)
Record Dates: First submitted 2022-05-31; First posted 2022-06-24 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Renal impairment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mild renal impaired subjects (Experimental): Administration of a single dose of CH6001 800 µg in mild renal impaired subjects.
  Interventions: Drug: CH6001
- Moderate renal impaired subjects (Experimental): Administration of a single dose of CH6001 800 µg in moderate renal impaired subjects.
  Interventions: Drug: CH6001
- Severe renal impaired subjects (Experimental): Administration of a single dose of CH6001 800 µg in severe renal impaired subjects.
  Interventions: Drug: CH6001
- Healthy volunteers (Experimental): Administration of a single dose of CH6001 800 µg in healthy volunteers.
  Interventions: Drug: CH6001

INTERVENTIONS:
Drug: CH6001 — CHF6001 will be administered using the NEXThaler® DPI device

SUMMARY:
The purpose of the study is to obtain pharmacokinetics, safety and tolerability data after single administrations of CHF6001 in subjects with mild, moderate and severe renal impairment as well as healthy volunteers under the same setting.

ELIGIBILITY:
Inclusion Criteria

All subjects:

1. Subject's written informed consent obtained prior to any study-related procedure;
2. Male and female subjects aged 40 to 80 years inclusive at screening;
3. Ability to understand the study procedures and the risks involved, and ability to be trained to use the inhalers correctly and to generate sufficient peak inspiratory flow (PIF, at least 40 L/min) using the In-Check device set as per NEXThaler® inhaler resistance;
4. Subjects must weigh at least 45kg for females and 50 kg for males to participate in the study, and must have a body mass index (BMI) within the range of 18 to 35 kg/m2 inclusive;
5. Non- or ex-smokers who smoked < 5 pack years (pack years = the number of cigarette packs per day times the number of years) and stopped smoking > 1 year prior to screening;
6. Oral body temperature < 37.5°C;
7. Mean values of triplicate recording of 12-lead digitised electrocardiogram (ECG) considered as normal (40 beats per min [bpm] ≤ heart rate [HR] ≤ 110 bpm, 120 ms ≤ PR interval [PR] ≤ 210 ms, QRS interval [QRS] ≤ 120 ms, QT interval corrected using Fridericia's formula [QTcF] ≤ 450 ms for males and QTcF ≤ 470 ms for females);
8. Lung function measurements within normal limits at screening: forced expiratory volume within the first second (FEV1) > 80% predicted and FEV1/Forced vital capacity (FVC) ratio > 0.70;
9. For female subjects:

   a. Women of child bearing potential (WOCBP) fulfilling one of the following criteria: i. WOCBP with fertile male partners: they and/or their partner must be willing to use at least an acceptable effective birth control method from the signature of the informed consent and until follow up contact; or ii. WOCBP with non-fertile male partners (contraception is not required in this case); b. Female subjects of non-childbearing potential defined as physiologically incapable of becoming pregnant. Tubal ligation or partial surgical interventions are not acceptable;

   Healthy subjects only:
10. Good mental and physical status, determined on the basis of the medical history and a general clinical examination;
11. Blood pressure within normal limits at screening and prior to study treatment administration: diastolic blood pressure (DBP) 40-89 mmHg and systolic blood pressure (SBP) 90-139 mmHg, extremes included;
12. Serum creatinine within the normal range and an eGFR ≥ 90 mL/min/1.73 m2 as determined by the MDRD equation;
13. Matched to at least one renal impaired subject enrolled in the study with respect to age (±10 years), gender, race and body weight (±15%);

    Renal impaired subjects only:
14. Good mental status, determined on the basis of the medical history and a general clinical examination;
15. Blood pressure at screening and prior to study treatment administration: DBP 40 100 mmHg and SBP 90 170 mmHg, extremes included;
16. Subjects must have a chronic stable renal disease based on the medical history, physical examination, and clinical laboratory results:

    1. "Chronic" is defined as > 6 months;
    2. "Stable" is defined as the absence of significant progression and/or deterioration of the renal disease for the past 12 weeks (fluctuations in creatinine levels within ±20% in the last 12 weeks are accepted); Subjects may have concurrent stable medical conditions in addition to renal impairment, but may be included only if the Investigator, in consultation with the Sponsor's Clinical Research Physician, considers that the condition will not introduce an additional risk factor, and will not interfere with the study objectives and procedures (e.g. subjects with stable diabetes or essential hypertension may be included);
17. Subjects with renal impairment must have the following absolute eGFR values as determined by the MDRD equation: mild renal impairment must have an absolute eGFR of ≥ 60 to < 90 mL/min/1.73 m2; moderate renal impairment must have an absolute eGFR of ≥ 30 to < 60 mL/min/1.73 m2; severe renal impairment must have an absolute eGFR of < 30 mL/min/1.73 m2 not requiring dialysis.

Exclusion Criteria

All subjects:

1. Participation to another clinical study where an investigational treatment was received, and last investigations were performed less than 8 weeks prior to screening;
2. Subjects with history of breathing problems (i.e. history of asthma including childhood asthma);
3. Positive human immunodeficiency virus (HIV) 1 or HIV2 serology;
4. Positive results from the Hepatitis serology which indicates acute or chronic hepatitis B or hepatitis C at screening (i.e. positive hepatitis B surface antigen [HBsAg], hepatitis B core antibody [immunoglobulin M antibody to hepatitis B core antigen, IgM anti-HBc], hepatitis C virus [HCV] antibody);
5. Documented coronavirus disease 2019 (COVID-19) diagnosis within the last 8 weeks, or complications from this disease, which have not resolved within 14 days prior to screening or to study treatment administration;
6. Blood donation or blood loss (≥ 450 mL) less than 2 months prior to screening or prior to study treatment administration;
7. Abnormal liver enzymes at screening (alanine aminotransferase [ALT] or Aspartate aminotransferase [AST] > 1.5 times the upper limit of normal [ULN], total bilirubin > 1.5 times the ULN);
8. Current haemodialysis or peritoneal dialysis or indications for these procedures;
9. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of orally administered drugs (e.g. history of bariatric surgery, stomach/intestinal significant resection, portacaval shunting);
10. Subject with severe heart failure as defined by the New York Heart Association functional classification III and IV;
11. Positive urine test for cotinine;
12. Documented history of alcohol abuse within 12 months prior to screening or a positive alcohol breath test;
13. Documented history of drug abuse within 12 months prior to screening or a positive urine drug screen evaluated at screening or prior to study drug administration;
14. Intake of non-permitted concomitant medications;
15. Presence of any current infection, or previous infection that resolved less than 7 days;
16. Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the study;
17. Unsuitable veins for repeated venepuncture;
18. Heavy caffeine drinker (average of > 5 cups or glasses per day of caffeinated beverages e.g. coffee, tea, cola, calculated by number of standard espresso portions);
19. For females only: pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive serum human chorionic gonadotropin laboratory test;
20. Contra-indications/warnings/precaution for use: contra indications to the investigational medicinal product (IMP) constitute an exclusion criterion;
21. The use of any kind of smoking electronic devices within 6 months before screening;

    Healthy subjects only:
22. Abnormal haemoglobin [Hb] level defined as < 130 g/L for males and < 110 g/L for females at screening;
23. Current diagnosis or history of nephrolithiasis (kidney stone);
24. Clinically relevant and uncontrolled respiratory, cardiovascular, hepatic, gastrointestinal, renal, endocrine, metabolic (especially subjects with deficiency in glucuronidation), neurologic, haematologic, neoplastic or psychiatric disorders that may interfere with successful completion of this study according to the Investigator's judgment;
25. Clinically relevant abnormal laboratory values at screening suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the subject or the evaluation of the result of the study according to the Investigator's judgment;

    Renal impaired subjects only:
26. Abnormal Hb level defined as ≤ 80 g/L at screening;
27. Clinically relevant and/or uncontrolled respiratory, cardiovascular, hepatic, gastrointestinal, endocrine, metabolic (especially subjects with deficiency in glucuronidation), neurologic, haematologic, neoplastic or psychiatric disorders that may interfere with successful completion of this study;
28. Acute renal disease caused by drug toxicity;
29. History of clinically significant (CS) chronic or recurrent urinary tract infection, active and requiring antibiotic treatment within the past 30 days;
30. Secondary renal disease associated with impaired liver metabolism (hepatorenal syndrome) or due to malignancy;
31. Significant risk factors for progression of the renal disease within 3 months prior to screening (e.g. uremic pericarditis, pleuritis, bleeding disorders, eGFR < 15 mL/min/m2);
32. Subjects who underwent a nephrectomy;
33. Subjects with a functioning organ transplant or who are registered on a transplant list.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC) of total plasma CHF6001 | Over 240 hours after CHF6001 administration
  Area under the plasma concentration versus time curve for total plasma CHF6001 after a single-dose of CHF6001
Maximum of Concentration (Cmax) of total plasma CHF6001 | Over 240 hours after CHF6001 administration
  Peak plasma concentration for total plasma CHF6001 after a single-dose of CHF6001

SECONDARY OUTCOMES:
Pharmacokinetic parameter ( Cmax) | Over 240 hours after administration in blood
  Peak Plasma Concentration (Cmax) for CHF6001 unbound plasma
Pharmacokinetic parameter (AUCt) | Over 240 hours after administration in blood
  Area under the plasma concentration versus time curve (AUCt) for CHF6001 unbound plasma
Pharmacokinetic parameter (AUC0-72) | Over 240 hours after administration in blood
  Area under plasma concentration from 0 to 72hours (AUC0-72) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (AUC0-240) | Over 240 hours after administration in blood
  Area under plasma concentration from 0 to 240hours (AUC0-240) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (AUC0-∞) | Over 240 hours after administration in blood
  Area under plasma concentration from 0 to infinity(AUC0-∞) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (tmax) | Over 240 hours after administration in blood
  Time of the maximum plasma concentration (tmax) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (t1/2) | Over 240 hours after administration in blood
  Terminal half-life (t1/2) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (CL/F) | Over 240 hours after administration in blood
  Apparent systemic clearance (CL/F) for CHF6001
Pharmacokinetic parameter (AUCt) | Over 240 hours after administration in blood
  Area under the plasma concentration versus time curve (AUCt) for CHF5956 and CHF6095
Pharmacokinetic parameter (Cmax) | Over 240 hours after administration in blood
  Peak Plasma Concentration (Cmax) for CHF5956 and CHF6095

CONTACTS AND LOCATIONS:
Locations (1):
- MC Comac Medical Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piccinno A, Pittelli MG, Balzano D, Rizzo E, Bellatti P, Rostello C, Emirova A. Evaluating the Impact of Hepatic or Renal Impairment on Tanimilast (CHF6001) Pharmacokinetics: Two Open-Label, Parallel-Group, Single-Center Studies. Clin Transl Sci. 2025 May;18(5):e70261. doi: 10.1111/cts.70261. PMID 40391696